CLINICAL TRIAL: NCT03353584
Title: Pain Management of Vaso-Occlusive Crisis in Children and Young Adults With Sickle Cell Disease-Effect of Virtual Reality Technology
Brief Title: Effect of Virtual Reality Technology for Pain Management of Vaso-Occlusive Crisis in Patients With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PMVOCVR
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: Virtual reality; Pain; Nonpharmacological
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Pain | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants receive standard care treatment for their vaso-occlusive crisis. Participants will be randomized by age.
- Virtual Reality (Active Comparator): Participants receive standard care treatment for their vaso-occlusive crisis. In addition, they will have a 15-minute Virtual Reality Therapy session. Participants will be randomized by age.
  Interventions: Other: Virtual Reality Therapy

INTERVENTIONS:
Other: Virtual Reality Therapy — The VR intervention consists of an interactive audio and visual underwater experience designed to serve as a calming distraction activity. The VR software (Kind VR® Aqua) was developed by KindVR specifically for the purpose of pain distraction in a hospital setting.
  Other Names: VR therapy
  Arms: Virtual Reality

SUMMARY:
Acute vaso-occlusive crisis (VOC) is the most common complication in patients with sickle cell disease (SCD) and pain related to VOC is often inadequately treated. This is a phase II randomized controlled clinical trial evaluating the efficacy of virtual reality technology when added to standard pain management for patients with sickle cell disease who are experiencing acute pain crisis in the ambulatory care setting. Patients will be randomized to receive either standard management only or standard management in addition to virtual reality therapy. The remainder of care for the painful event will continue per institutional standards according to clinical indication, including reassessment and documentation of pain and additional doses of pain medicines by intravenous (IV) or oral route. Pain scores and opioid requirement will be measured and compared across treatment arms, along with the outcomes of discharge from clinic versus admission to the inpatient unit.

PRIMARY OBJECTIVE: To assess the efficacy of virtual reality (VR) technology in reducing pain at 30 minutes after intervention during an acute vaso-occlusive crisis in patients with sickle cell disease. Primary endpoint will be change in pain scores in Standard versus VR arms, between the first pain assessment at the time of presentation and the subsequent pain assessments up to 30 minutes after intervention.

Secondary Objectives:

* To compare total opioid consumption from the time of presentation to the time of discharge from acute care setting in Standard versus VR arms.
* To assess the efficacy of virtual reality (VR) technology in reducing pain at 60 minutes after the first IV medication administered or 60 minutes after completion VR during an acute vaso-occlusive crisis in patients with sickle cell disease.

DETAILED DESCRIPTION:
After consenting to participate in this study, patients will be randomized to receive either standard care therapy for VOC or to receive standard care therapy plus a 15-minute virtual reality (VR) session. They will be additionally randomized into strata by age: 6 to 11 years, 12 to 18 years, and 19 to 25 years. At the end of therapy or therapy plus the VR session, they will be asked to complete a 5-minute satisfaction survey. Information will also be collected from the medical record about the pain episode, including pain scores, medicines used, and time needed for pain to lessen.

Standard care for management of an acute VOC includes parenteral hydration and pain management with non-steroidal anti-inflammatory agents, such as Toradol or Ibuprofen, and opioids. Pain scores will be measured at three different time points: baseline at presentation, at 30±10 minutes after first intravenous (IV) analgesic medication, and at 60±10 minutes after first IV analgesic medication.

Use of VR will be included in addition to the standard care for management of patients randomized to VR arm. VR is an interactive technology that allows the user to interface with a three dimensional computer-generated environment by means of a lightweight head mounted display. The user is transported into a relaxing VR environment that diverts their attention away from pain. The duration of VR session is 15 minutes. Pain scores will be measured at three different time points: baseline at presentation, at 15±10 minutes after completion of VR therapy, and at 60±10 minutes after completion of VR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have sickle cell disease (any genotype), documented in the St. Jude medical record.
* Participant must be seeking care for acute VOC pain at St. Jude Children's Research Hospital.
* Participant age must be ≥ 6 years and ≤ 25 years.
* English speaking

Exclusion Criteria:

* Prior randomization in this study.
* Patients are currently enrolled on another pain management interventional trial for the presenting pain crisis.
* Mild pain (score <4), or pain for which treatment with opioid is not indicated.
* Pain in combination with other clinical symptoms that require additional interventions, including fever with focus, acute chest syndrome, acute injury, or splenic sequestration.
* Developmental or psychiatric disorders like autism, claustrophobia or other disabilities like vision and hearing defects etc. that preclude the use of a head mounted device.
* Inability or unwillingness of research participant or legal guardian/ representative to give written informed consent.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | Baseline and up to 30 minutes after intervention
  The highest pain score based on all scores at different body pain locations is used as the pain score. The changes in pain scores in two arms between baseline and 30 minutes post study intervention will be summarized and compared using Wilcoxon rank sum test at a significance level of 0.1.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Methodist Comprehensive Sickle Cell Center, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols